CLINICAL TRIAL: NCT06395077
Title: Diagnostic Efficiency of Low-dose Cone-beam Computed Tomography in Post-graft Evaluation of Swedish Paediatric Patients With Alveolar Clefts
Brief Title: Diagnostic Efficiency of Low-dose Cone-beam Computed Tomography in Post-graft Evaluation.
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Kristina Hellén-Halme, Professor, Malmö University
Other Study IDs: FO 2020/401
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Alveolar Cleft
Keywords: CBCT; Low-dose; Alveolar cleft

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBCT low-dose protocol — The patient underwent two CBCT examinations (Accuitomo 170; J Morita Corp., Kyoto, Japan): one examination followed the clinical standard-dose protocol (exposure settings: 90 kV, 5 mA, and 9.4 s), and one, the low-dose protocol (90 kV, 2 mA, 9.4 s).

SUMMARY:
Evaluation of a Low-dose exposure CBCT protocol for post-graft evaluation of treatment of cleft patients

DETAILED DESCRIPTION:
The patient underwent two CBCT examinations (Accuitomo 170; J Morita Corp., Kyoto, Japan): one examination followed the clinical standard-dose protocol (exposure settings: 90 kV, 5 mA, and 9.4 s), and one, the low-dose protocol (90 kV, 2 mA, 9.4 s). The field of view (FOV) was 6.0 cm x 6.0 cm, the rotation mode was 180 degrees, and voxel size was 0.125 mm. Volume was reconstructed in slices of 1-mm thickness and interval. The dose area products (DAP) were 423 mGy cm2 for the clinical, standard-dose protocol and 172 mGy cm2 for the low-dose protocol.

The aim was to establish if a low-dose protocol could provide diagnostically acceptable image quality for assessing bone healing after alveolar bone grafting.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral facial clefts who had undergone alveoalar bone grafting. Healing control after 6 months.

Exclusion Criteria:

-

Ages: 7 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: patients with oral facial clefts who had undergone alveoalar bone grafting. Healing control after 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of post grafting in patients with clefts. | 2 years
  CBCT investigation after surgery of patients with alveolar clefts.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Hellén-Halme, Principal Investigator — Malmo university
Locations (1):
- Kristina Hellen-Halme, Malmo, Sweden

REFERENCES:
- [Derived] Vicente A, Cederhag J, Rashidi N, Wiedel AP, Becker M, Brogardh-Roth S, Shi XQ, Hellen-Halme K. Low-Dose Cone-Beam Computed Tomography in Swedish Pediatric Patients With Alveolar Clefts Following Alveolar Bone Grafting-A Clinical Study. Clin Exp Dent Res. 2024 Dec;10(6):e70021. doi: 10.1002/cre2.70021. PMID 39497332